CLINICAL TRIAL: NCT04291079
Title: A Phase 1, Open-Label, Dose-Escalation, and Dose-Expansion Study to Investigate the Safety, Tolerability, PK, PD, and Efficacy of SRK-181 Alone and in Combination With Anti-PD-(L)1 Antibody Therapy in Patients With Locally Advanced or Metastatic Solid Tumors (DRAGON)
Brief Title: SRK-181 Alone or in Combination With Anti-PD-(L)1 Antibody Therapy in Patients With Locally Advanced or Metastatic Solid Tumors (DRAGON)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scholar Rock, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRK-181-001
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: Solid Tumor; Metastatic; Melanoma; Urothelial; Non-Small Cell Lung Carcinoma; ccRCC; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — SRK-181

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A1: Dose Escalation (Experimental): Part A1 determined the maximum tolerated dose (MTD) or maximum administered dose (MAD) of SRK-181 as a single agent and the recommended Phase 2 dose (RP2D) of SRK-181 as a single-agent.
  Interventions: Biological: SRK-181
- Part A2: Dose Escalation (Experimental): Part A2 determined the MTD or MAD of SRK-181 in combination with anti-PD-(L)1 antibody therapy and the RP2D of SRK-181 in combination with anti-PD-(L)1 antibody therapy for use in Part B.
  Interventions: Biological: SRK-181; Biological: anti-PD-(L)1 antibody therapy
- Part B: Dose Expansion (Experimental): In Part B, parallel cohorts of patients with Non-Small Cell Lung Cancer (NSCLC), Urothelial Carcinoma (UC), Cutaneous Melanoma (MEL), Clear Cell Renal Cell Carcinoma (ccRCC), Head and Neck Squamous Cell Carcinoma (HNSCC), or other advanced or metastatic solid tumor type that is not NSCLC, UC, MEL, or ccRCC were enrolled to confirm the tolerability of the RP2D of SRK-181 (determined in Part A2) and to evaluate the anti-tumor activity of SRK-181 in combination with an anti-PD-(L)1 antibody therapy.
  Interventions: Biological: SRK-181; Biological: anti-PD-(L)1 antibody therapy
- Long Term Extension Phase (LTEP) (Experimental): Patients may continue treatment in a LTEP:
  * Part A1: Patients may continue treatment with SRK-181 as a single agent at the RP2D in the LTEP following 3 cycles of treatment with SRK-181 as a single agent in Part A1.
  * Part A2: Patients may continue treatment with SRK-181 at the RP2D in combination with anti-PD-(L)1 antibody therapy in the LTEP following 3 cycles of treatment with SRK-181 in combination with anti-PD-(L)1 antibody therapy in Part A2.
  * Part B: Patients may continue treatment with SRK-181 in combination with anti-PD-(L)1 antibody therapy following 9 cycles of treatment with SRK-181 in combination with anti-PD-(L)1 antibody therapy in Part B
  Interventions: Biological: SRK-181; Biological: anti-PD-(L)1 antibody therapy

INTERVENTIONS:
Biological: SRK-181 — anti-latent TGFβ1 monoclonal antibody
Biological: anti-PD-(L)1 antibody therapy — approved anti-PD-(L)1 antibody therapy for each tumor type
  Arms: Long Term Extension Phase (LTEP); Part A2: Dose Escalation; Part B: Dose Expansion

SUMMARY:
This was a multi-center, open-label, Phase 1, first-in-human (FIH), dose-escalation, and dose expansion study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of SRK-181 administered alone and in combination with anti-PD-(L)1 therapy in adult patients with locally advanced or metastatic solid tumors. The study was divided into 3 treatment parts (Part A1, Part A2, and Part B) and a Long-Term Extension Phase (LTEP).

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has a histologically documented solid tumor that is metastatic or locally advanced, for which SoC therapy does not exist, has failed in the patient, or is not tolerated by the patient, or for which the patient has been assessed by the Investigator as not being a suitable candidate or otherwise ineligible for the SoC therapy.
* For Part A2:

  o Patient must have a history of anti-PD-(L)1 antibody nonresponse presenting (based upon the Investigator's assessment) either as progressive disease or stable disease (e.g., not improving, but also not worsening, clinically or radiographically) after at least 3 cycles of treatment with the most recent anti-PD-(L)1 antibody therapy (alone or in combination with chemotherapy) approved for that tumor type. (Note: if the duration of prior anti-PD-1 therapy is shorter than 3 cycles and the reason for discontinuation is progressive disease, the progression should be associated with clinical deterioration.)
* For Part B Cohort NSCLC, UC, MEL and ccRCC:

  * Patient must be diagnosed with one of the following disease-specific solid tumors of NSCLC, UC, or MEL, and must have a history of primary nonresponse to anti-PD-1 therapy (alone or in combination with other therapy), presenting the best response (based upon the Investigator's assessment) either as progressive disease or stable disease (e.g., not improving, but also not worsening, clinically or radiographically) after at least 3 cycles of treatment.
  * For Cohort NSCLC, patients who have genomic tumor aberrations for which a targeted therapy is available (e.g., anaplastic lymphoma kinase, EGFR) must have progressed on an approved therapy for these aberrations or did not tolerate an approved therapy for these aberrations, or were not considered suitable candidates/ were otherwise ineligible for an approved therapy for these aberrations.
  * For Cohort ccRCC, patients must have a histologically confirmed diagnosis of RCC with a predominant clear cell component and must have received at least 1 prior line of anti-PD-1 treatment (alone or in combination with other therapy) and have had disease progression clinically or radiographically on the most recent anti-PD-1 treatment
  * Up to 3 lines of treatment are allowed between the last dose of anti-PD-1 and enrollment.
* For Part B Cohort HNSCC:

  * Patients must have a histologically confirmed diagnosis of recurrent or metastatic HNSCC that is non-amendable to curative therapy (e.g., radiation or surgery).
  * The primary tumor location must be the oropharynx, oral cavity, hypopharynx, or larynx. Primary tumor site of nasopharynx (any histology) or unknown primary tumor are not eligible.
  * Patients must have received one prior line of anti-PD-1 treatment (alone or in combination with other therapy) and have had disease progression clinically or radiographically on the anti-PD-1 treatment.
  * Up to one line of treatment are allowed between the last dose of anti-PD-1 and enrollment.
  * For patients with primary oropharyngeal cancer, patients must have results from testing of human papillomavirus (HPV) or P16 status.
* For Part B Cohort Any Other (enrollment complete): Patient must be diagnosed with any other solid tumor type that is not NSCLC, UC, MEL, or ccRCC for which the patient has had a history of primary anti PD (L)1 antibody nonresponse, presenting the best response (based upon the Investigator's assessment) as progressive disease, after prior anti-PD-(L)1 antibody therapy (alone or in combination with other therapy) currently approved for that tumor indication
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed at Screening.
* Patient must have an Eastern Cooperative Oncology Group performance status (PS) 0-1.
* Patient must have a predicted life expectancy of ≥ 3 months.
* Women of child-bearing potential (WOCBP) must have a negative urine or serum pregnancy test up to 24 hours prior to first dose of SRK-181.
* WOCBP and males with female partners of childbearing potential must agree to use adequate birth control throughout their participation and for 90 days following the last dose of SRK-181.

Key Exclusion Criteria:

* For Part A1 only:

  * Patient has had anti-PD-(L)1 antibody therapy ≤ 28 days prior to the first dose of SRK-181.
  * Patient is receiving concurrent anti-cancer treatment, including anti-PD-(L)1 antibody therapy, either approved or investigational, within 28 days prior to the first dose of SRK-181.
* For Part A2 and Part B only:

  * Patient is receiving concurrent anti-cancer treatment, with the exception of an anti-PD-(L)1 antibody therapy for Part A2 or Part B, either approved or investigational, within 28 days prior to the first dose of SRK-181.
  * Patient has received biologic therapy (except for anti-PD-(L)1 antibody therapy for Part A2 or Part B), <28 days prior to the first dose of SRK-181.
  * Patient has received systemic cytotoxic chemotherapy (except for in combination with anti-PD-(L)1 antibody therapy) <28 days prior to the first dose of SRK-181.
  * Patient has received targeted small molecule therapy within 5 half-lives of the compound prior to the first dose of SRK-181.
  * Patient has a history of intolerance or treatment discontinuation due to severe irAE or other adverse reaction from prior anti-PD-(L)1 antibody therapy.
* Patient has a hypersensitivity to anti-PD-(L)1 antibody therapy.
* Patient has the documented presence of neutralizing ADA to anti-PD-(L)1 antibody therapy.
* Patient has a diagnosis of immunodeficiency, either primary or acquired.
* Patient is symptomatic or has uncontrolled brain metastases, leptomeningeal disease, or spinal cord compression not definitively treated with surgery or radiation.
* Patient has current second malignancy at other sites (exceptions: adequately treated in situ carcinoma [e.g., cervical], non-MEL skin cancer, bilateral synchronous discordant breast cancer, or indolent prostate cancer under observation). A past history of other malignancies is allowed as long as patient has been free of recurrence for ≥ 2 years, or if the patient has been treated with curative intent within the past 2 years and, in the opinion of the Investigator, is unlikely to have a recurrence.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single agent SRK-181 | The first 21 days of study treatment
  Dose limiting toxicities (DLTs), as assessed by the Investigator, but not including toxicities clearly related to disease progression or intercurrent illness
Safety and tolerability of SRK-181 in combination with anti-PD-(L)1 antibody therapy | The first 21 days of study treatment
  Dose limiting toxicities (DLTs), as assessed by the Investigator, but not including toxicities clearly related to disease progression or intercurrent illness

SECONDARY OUTCOMES:
PK of SRK-181 alone and in combination with anti-PD-(L)1 antibody therapy | Cycle 1 and Cycle 3 (each cycle is 21 days)
  Maximum drug concentration (Cmax)
PK of SRK-181 alone and in combination with anti-PD-(L)1 antibody therapy | Cycle 1 and Cycle 3 (each cycle is 21 days)
  Time to Cmax (Tmax)
PK of SRK-181 alone and in combination with anti-PD-(L)1 antibody therapy | Cycle 1 and Cycle 3 (each cycle is 21 days)
  Last validated plasma concentration (Clast)
PK of SRK-181 alone and in combination with anti-PD-(L)1 antibody therapy | Cycle 1 and Cycle 3 (each cycle is 21 days)
  Time to Clast (Tlast)
PK of SRK-181 alone and in combination with anti-PD-(L)1 antibody therapy | Cycle 1 and Cycle 3 (each cycle is 21 days)
  Half-life (t1/2)
Anti-tumor activity of SRK-181, alone or in combination wit anti-PD-(L)1 antibody therapy as potential indicators of clinical response | 6 months
  Objective response, defined as a CR or PR, as determined by RECIST v1.1 or iRECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Lu Gan, MD, Study Director — Scholar Rock, Inc.
Locations (22):
- United States (18):
  - St. Jude Crosson Cancer Institute, Fullerton, California
  - University of California - San Diego, La Jolla, California
  - The Oncology Institute, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Advent Health, Celebration, Florida
  - Memorial Cancer Institute - South Broward Hospital District, Hollywood, Florida
  - H. Lee Moffitt Cancer Center& Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Tennessee Oncology, Sarah Cannon Research Institute, Nashville, Tennessee
  - BUMC Mary Crowley Cancer Research Centers, Dallas, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- South Korea (4):
  - Korea University Ansan Hospital, Ansan-si
  - Seoul National University - Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yap TA, Sweis RF, Vaishampayan U, Kilari D, Gainor JF, McKean M, Barve M, Tarhini AA, Bockorny B, Sonpavde G, Park D, Babu S, Ju Y, Liu L, Henry S, Tirucherai GS, DeWall S, Qatanani M, Marantz JL, Gan L. Linavonkibart and pembrolizumab in immune checkpoint blockade-resistant advanced solid tumors: a phase 1 trial. Nat Med. 2026 Jan 13. doi: 10.1038/s41591-025-04157-w. Online ahead of print. PMID 41530380